CLINICAL TRIAL: NCT05634928
Title: Construction of a Database for Thrombotic Microangiopathy
Brief Title: Construction of a Database for TMA
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: SOOCHOW-HY-2022-13
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Thrombotic Microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMA: TMA patients
  Interventions: Other: collection data

INTERVENTIONS:
Other: collection data — collection data

SUMMARY:
Information about patients was collected by reviewing the Hitech case system and telephone and outpatient follow-up, and the case database was constructed by Epidata software. The sample size is expected to be 200 cases, the participating hospital is the First Affiliated Hospital of Soochow University, and the study time frame is from Dec 1, 2022, to Nov 31, 2027. The observation indexes of the study include the basic information of patients' age and gender and the clinical-related data of thrombotic microangiopathy.

ELIGIBILITY:
Inclusion Criteria:

* The patient has elevated lactate dehydrogenase to more than twice the baseline value, platelets less than 20 or decreased by more than 50% within 24 hours, and more than 2% of schistocytes visible on a peripheral blood smear. Alternatively, pathological sections show extensive micro thrombosis.

Exclusion Criteria:

* The investigator considers the subject unable or unwilling to cooperate with the study procedures.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 500 eligible TMA patients are to be collected for this project.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with stroke | 5 years from the time of entering the database.
  Stroke was assessed with MRI imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China